CLINICAL TRIAL: NCT06962306
Title: Perioperative Methadone Use for Cleft Palate Repair: A Randomized Controlled Trial
Brief Title: Optimizing Perioperative Analgesia to Lower Pain Following Cleft Palate Surgery
Acronym: OPAL-Cleft
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00117598
Record Dates: First submitted 2025-04-30; First posted 2025-05-08 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-04

CONDITIONS: Cleft Palate; Pain; Postoperative Care; Perioperative Care; Children
Keywords: Cleft palate surgery; Perioperative pain management; Analgesia; Methadone
MeSH Terms: conditions — Cleft Palate; Pain; Agnosia | interventions — Methadone; Fentanyl; Hydromorphone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Methadone (Active Comparator): Methadone 0.2-0.25 mg/kg actual body weight
  Interventions: Drug: Methadone hydrochloride
- Fentanyl/Hydromorphone (Active Comparator): Fentanyl/Hydromorphone per routine care
  Interventions: Drug: Fentanyl/Hydromorphone

INTERVENTIONS:
Drug: Methadone hydrochloride — Initial dosing 0.2mg/kg, potential to escalate to 0.25mg/kg following interim analysis
  Arms: Methadone
Drug: Fentanyl/Hydromorphone — Per routine care
  Arms: Fentanyl/Hydromorphone

SUMMARY:
The purpose of this study is to compare the use of short acting opioids (fentanyl/hydromorphone) with long acting opioids (methadone) for pain control following cleft palate surgery in infants and young children.

DETAILED DESCRIPTION:
This is a single center, randomized, double blind, parallel-group dose escalation investigation in infants and children undergoing cleft palate surgery which will compare post operative pain control indices for patients receiving short acting versus long acting opioids as perioperative analgesics. Surgical and anesthesia care, except for opioid management, are not altered for study purposes. Subjects are randomized 2:1 to either long-duration (methadone) or short-duration opioid (fentanyl, hydromorphone) through the perioperative period. Exploratory data will be collected for up to 30 days post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 months to 4 years of age
* Primary cleft palate repair
* Signed informed consent by parent or legal guardian

Exclusion Criteria:

* History of chronic kidney or liver disease
* Planned admission to the Pediatric Intensive Care Unit (PICU)
* Additional procedures under general anesthesia for which opioids would be prescribed
* Any patient ineligible for study participation at the discretion of the investigators

Ages: 6 Months to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2027-06-04 (Estimated); Study Completion 2027-07-04 (Estimated)

PRIMARY OUTCOMES:
Total amount of opioids medication administered | From PACU discharge through postoperative day 1 (POD1)
  Post-PACU in-hospital opioid use in oral morphine milligram equivalents (OMEs) per kilogram through POD1

SECONDARY OUTCOMES:
Total amount of opioid medications administered | Up to 7 days after surgery
  Total (post-PACU in-hospital and post-discharge) opioids used (number of daily doses and OME/kg)
Postanesthesia Care Unit (PACU) opioid medication administration | Up to 6 hours after surgery
  Binary (yes/no) need for opioid administration in the PACU
Area under the curve (AUC) pain trajectories | Through hospital discharge (up to 4 days)
  In-hospital AUC pain trajectories calculated from pain intensity scores on the Face, Legs, Activity, Cry, Consolability (FLACC) pain scale. The FLACC pain scale has a range of 0 to 10, where 0=no pain and 10=worst possible pain.
Average daily pain intensity | Up to 7 days after surgery
  Average daily pain scores using the Face, Legs, Activity, Cry, Consolability (FLACC) pain scale. The FLACC pain scale has a range of 0 to 10, where 0=no pain and 10=worst possible pain.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M. Einhorn, M.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared at the discretion of the PI upon reasonable request.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: IPD will be available 1 year after study completion.